CLINICAL TRIAL: NCT03934164
Title: MAESTRO: Molecular Stratification Profiling Protocol in Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Molecular Stratification Profiling Protocol in Metastatic Castration Resistant Prostate Cancer (mCRPC) - MAESTRO
Acronym: MAESTRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Prostate Cancer UK (Other)
Responsible Party: Sponsor
Other Study IDs: ICR-CTSU/2016/10059
Record Dates: First submitted 2018-12-21; First posted 2019-05-01 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Prostate Cancer; Castration-resistant Prostate Cancer
Keywords: prostate; molecular stratification
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, observational, molecular stratification profiling study. Patients with mCRPC who have received at least one standard treatment for mCRPC will be approached to participate in MAESTRO. Patients must have archival tumour available and be willing to undergo a fresh tumour biopsy for molecular analyses. Tumour tissue (archival and fresh), research blood samples and saliva will be sent to the central laboratory for analysis to identify molecular aberrations through targeted or broader molecular analyses (e.g. exome, transcriptome) and orthogonal assays (e.g. immunohistochemistry; digital droplet PCR). When the results are available, depending on patients choice, the results will be discussed. If significant results are indicated, patients will be recommended to have follow up with a cancer geneticist to discuss the implications of these results for their personal and family's health.

There is a safety follow up 30 days after collection of study biopsy or blood samples. Patients will also be followed up for overall survival and subsequent anticancer treatment every 6 monthly via medical notes or telephone calls.

DETAILED DESCRIPTION:
This study is a prospective, observational, molecular stratification profiling study.

mCRPC patients who have received at least one standard treatment for mCRPC will be approached to participate in MAESTRO. Patients must have archival tumour available and be willing to undergo a fresh tumour biopsy for molecular analyses. Following consent to MAESTRO, tumour tissue (archival and fresh), along with the research blood samples and saliva sample will be sent to the central laboratory for analysis to identify molecular aberrations through targeted or broader genomic analyses (e.g. exome, transcriptome) and orthogonal assays (e.g. immunohistochemistry; digital droplet PCR).

Patients will not receive any treatment as part of MAESTRO. Results of the molecular characterisation will be provided to the treating investigator to be fed back to the patient, depending on patient's choice on disclosing the results.

The following research samples are collected under as part of this study:

* Where available, excess archival tumour tissue from previous biopsies or routine surgical procedures will be retrospectively collected.
* Fresh tissue specimens will be obtained for patients who are undergoing standard of care interventions OR patient will undergo a bone marrow biopsy or an ultrasound /CT guided tumour biopsy of a safely accessible lesion. Fresh tumour specimens will be processed and/or frozen.
* Sequencing analysis of tissues will be done and results will be made available in real time. Clinically significant results will be disclosed to patients and their clinicians as per patient consent.
* Research samples for blood, serum, plasma and saliva will be collected at the time of the biopsy.

Patients who elected (optional consent) to receive sequencing results regarding incidental clinically significant findings, will be referred for genetic counselling.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged ≥18 years.
2. Histologically confirmed metastatic castrate resistant adenocarcinoma of the prostate
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 - 2.
4. Surgically or medically castrated, with testosterone levels of <50 ng/dL (<2.0 nM).
5. Confirmed metastatic disease on imaging.
6. Patients with tumour deemed by the designated investigator as safely suitable for fresh biopsy AND who are medically fit (according to local practice) to undergo a biopsy or procedure to acquire tumour tissue AND previously collected tumour specimens from prior surgery or biopsy available for analyses. An mCRPC biopsy collected within 6-months of trial entry can be used instead of this fresh biopsy if available and passes laboratory quality control requirements.
7. Willing and able to comply with the requirements of the sample collection including fresh tumour biopsy.
8. The subject is capable of understanding and complying with the protocol requirements and has given written informed consent.

Exclusion Criteria:

1. The presence of any haematological disorders, including coagulation disorders, which would be a contraindication if patient were to undergo a biopsy.
2. Any psychiatric illness/social situations that would limit compliance with study requirements.
3. Presence of any concurrent condition or situation, which, in the investigators opinion, may put the patient at significant risk, may confound the study results or may interfere significantly with the patient's participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from participating sites in the UK. Potential participants will be identified and discussed in oncology clinics and Multi-Disciplinary Team (MDT) meetings.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Number of molecular aberrations in diagnostic archive and fresh mCRPC tissue | 4-6 weeks
  The prevalence of molecular aberrations in diagnostic archive and fresh mCRPC will be calculated with 95% confidence intervals.

SECONDARY OUTCOMES:
Quantify the association between molecular aberrations and baseline prognostic characteristics | 4-6 weeks
  The association between identified molecular aberrations and baseline characteristics, known to be prognostic factors, will be quantified. Associations will be determined using Fisher's exact test for categorical characteristics and for continuous characteristics either a Wilcoxon rank sum test or t test will be used depending on the results of normality testing.
Changes in molecular aberrations | 4-6 weeks
  Changes in the molecular features of tumour biopsies acquired at diagnosis and fresh mCRPC will be quantified to demonstrate any differences in the molecular aberrations within the same patient's tumour.
Safety - Review of biopsy-related adverse events: occurrence of at least one grade 3 or 4 event | 30 days after study biopsy/blood collection
  All events experienced by patients related to study procedures (collection of a fresh biopsy or blood samples) will be recorded and graded using CTCAE version 5 criteria and specifically the occurrence of at least one grade 3 or 4 event. Adverse events will be summarised by grade according to the worst grade experienced. In addition, the most frequently observed AEs will be summarised. The overall proportion of patients experiencing at least one grade 3 or 4 event will be presented by study procedure.
Time to development of CRPC | From the date of diagnosis to the date of confirmed mCRPC, through study completion, up to 5 years
  This is defined in whole days as the time from the date of diagnosis to the date of confirmed CRPC. The median time and interquartile range will be determined per molecular aberration. Analyses will be conducted per molecular aberration and will use the Kaplan-Meier method and Cox proportional hazard models. Analyses will adjust for known baseline characteristics and previous treatments received using multivariable Cox proportional hazard models.
Overall Survival (OS) | From the date of confirmed CRPC to the date of death from any cause, , through study completion, up to 5 years
  OS will be measured from the date of CRPC to the date of death (whatever the cause). Survival time of living patients will be censored on the last date a patient is known to be alive or lost to follow-up. Analyses will use the Kaplan Meier method and Cox proportional hazard models by molecular aberration. Multivariable Cox proportional hazard models will include established prognostic factors such as site of disease.

OTHER OUTCOMES:
Circulating Free DNA | 4-6 weeks
  To evaluate the agreement between molecular aberrations found in cfDNA and tumour biopsies (fresh and archival) from primary (prostate) or metastatic site. Agreement will be determined per paired sample for each molecular aberration using Cohen's kappa coefficient.
Circulating Tumour Cells | 4-6 weeks
  To acquire DNA from pure CTCs. To evaluate the agreement between molecular aberrations found in CTCs and tumour biopsies (fresh and archival) from primary (prostate) or metastatic site. Agreement will be determined per paired sample for each molecular aberration using Cohen's kappa coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, Principal Investigator — The Institute of Cancer Research and The Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHSFT, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided